CLINICAL TRIAL: NCT04922086
Title: The Effectiveness of Digital Planning and Guided Dual Technique in Aesthetic Crown Lengthening: A Randomized Controlled Clinical Trial
Brief Title: Digital Planning and Guided Dual Technique in Aesthetic Crown Lengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACL - UNIFAL
Record Dates: First submitted 2021-05-14; First posted 2021-06-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Tooth Eruption Disorder
Keywords: Crown Lengthening; Altered passive eruption; Gingival smile

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Patients will be submitted to ACL planned using cone beam computed tomography (CBCT), digital planning and guided dual technique.
  Interventions: Procedure: Guided dual aesthetic crown lengthening surgery
- Control group (Active Comparator): Patients will be submitted to the conventional ACL planned using clinical examination.
  Interventions: Procedure: Conventional aesthetic crown lengthening surgery

INTERVENTIONS:
Procedure: Conventional aesthetic crown lengthening surgery — The demarcation of the gingival zenith final position will be done on the teeth using a periodontal probe. This demarcation will be done through visual examination based on the crown length/width ratio and the position of the cemento-enamel junction (CEJ). The gingival margin of the central and canine incisors will be positioned at similar heights and a more coronal gingival contour will be determined for the lateral incisors. An internal bevel incision will be made with a blade on each tooth, preserving the interdental papillae. The incised gingival tissue will be removed using a periodontal curette in both groups. An internal bevel incision will be made in the involved teeth and a full thickness flap will be displaced up to the the mucogingival junction level to expose the bone crest (BC). Carbide drills and manual chisels will be used for bone resection to obtained a CEJ-BC distance of 3 mm. Simple interproximal interrupted sutures will be performed.
  Arms: Control group
Procedure: Guided dual aesthetic crown lengthening surgery — The double guide will be positioned and an internal bevel incision on each tooth will be made following the guide demarcation. After the initial incision, the incised gingival tissue will be removed using a periodontal curette. An internal bevel incision will be made in the involved teeth and a full thickness flap will be displaced up to the the mucogingival junction level to expose the bone crest (BC). The dual guide will be positioned again and the bone tissue will be removed using carbide drills and manual chisels following the double guide. No interproximal crestal bone will be removed. Simple interproximal interrupted sutures will be performed to stabilize the flap.
  Arms: Test group

SUMMARY:
Excessive gingival exposure, commonly named gingival smile, results in a dentogingival disharmony. One of the gingival smile treatment is the aesthetics-related crown lengthening surgery (ACL) to provide a adequate clinical crown length and diminish gingival display. In this context, digital planning and guided dual technique have been proposed to increase the effectiveness and predictability of the ACL. In this technique, an facial and dental analysis of the patient is performed and transferred to a digital model obtained by intraoral digital scan. The digital model is used to create a double guide that will determine the final position of the gingival and alveolar margin in the ACL. Despite the technique showing promising results, clinical studies evaluating the effectiveness of this technique are scarce. The present study aims to evaluate the digital planning and guided dual technique in the ACL in comparison to conventional technique in relation to the predictability/stability of the gingival margin positioning and patient satisfaction after the ACL. Twenty-four patients diagnosed with altered passive eruption type I subcategory B will be selected and divided into two groups. In the control group (n = 12) patients will be submitted to the conventional ACL planned using clinical examination; in the test group (n = 12) patients will be submitted to ACL using cone beam computed tomography (CBCT), digital planning and guided dual technique. Periodontal clinical parameters including probing depth (PS), clinical attachment level (CAL), clinical crown length (CCL), anatomical crown length (ACL) and cemento-enamel junction to alveolar bone crest distance will be evaluated clinically at baseline, in the immediate postoperative, 4, 8 and 12 months after the procedure. Participants will be submitted to questionnaires to assess satisfaction with the smile, gum and tooth characteristics and experience with the procedure. The investigators aim to demonstrate with the study the effectiveness of the both techniques and evaluate the clinical cost benefit for the patient and the dentist of the guided dual technique in relation to the conventional ACL technique.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers;
* Periodontal and systemically healthy;
* Patients with more than 20 teeth including the six maxillary anterior teeth;
* Altered passive eruption diagnosis (classified as type I subcategory B) in the quadratic anterior teeth.

Exclusion Criteria:

* Orthodontic treatment;
* Presence of prosthetic crowns;
* Extensive restorations;
* Extensive incisal edge attrition;
* Misalignment on maxillary anterior teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change of clinical crown length. | Baseline, immediately after the intervention, 4, 8 and 12 months.
  Measured as the distance between incisal edge and gingival marginal using a periodontal probe and its will determine the stability of the gingival margin in the both groups. The clinical crown length will be also measured using a cone beam computed tomography (CBCT)

SECONDARY OUTCOMES:
Change of gingival display. | Baseline, 4, 8 and 12 months.
  Measured as the distance between central incisor gingival margin during active smile and the inferior border of the upper lip vermilion using a periodontal probe.
Change of gingival width. | Baseline, immediately after the intervention, 4, 8 and 12 months.
  Measured as the distance between mucogingival junction and gingival margin, using the visual method.
Change of gingival margin position. | Baseline, 4, 8 and 12 months.
  Measured as the cemento-enamel junction to gingival margin distance using a periodontal probe.
Change of gingival thickness. | Baseline.
  Measured at the 3mm apical of gingival margin with a endodontics file inserted perpendicular to the surface until firm resistance was met, and recorded to the nearest millimetre using a digital caliber. The gingival thickness will be also measured using a cone beam computed tomography (CBCT).
Change of anatomic crown length. | During the intervention.
  Measured after flap elevation as the distance between incisal edge and cemento-enamel junction, along the long axis of the tooth using a periodontal probe and cone beam computed tomography (CBCT).
Distance between cemento-enamel junction and bone crest. | During the intervention.
  Measured of the distance between cemento-enamel junction and bone crest using a periodontal probe and cone beam computed tomography (CBCT).
Change of probing depth. | Baseline, 4, 8 and 12 months.
  Measured as the distance between gingival margin and bottom of the gingival sulcus using a periodontal probe.
Change of clinical attachment level | Baseline, 4, 8 and 12 months.
  Measured as the distance between cemento-enamel junction and bottom of the sulcus using a periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Suzane C Pigossi, PhD, Principal Investigator — Universidade Federal de Alfenas
Locations (1):
- Universidade Federal de Alfenas, Alfenas, Minas Gerais, Brazil